CLINICAL TRIAL: NCT06242106
Title: Effects of Self-stretching With and Without Aerobic Exercise on Glycemic Control, Fatigue and Stress in Gestational Diabetes
Brief Title: Effects of Self-stretching and Aerobic Exercise in Gestational Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S22C14G92006
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Gestational Diabetes
Keywords: Aerobic exercise,; Fatigue; Stress; Gestational diabetes; Glycemic control; Self-stretching
MeSH Terms: conditions — Diabetes, Gestational; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercises + self-stretching (Experimental): • After the baseline assessment, the patient in the experimental group received self-stretching with aerobic exercises. Self-stretching that includes butterfly stretch, wall stretching and cat and cow pose for 5 sec each and 10 repetitions, with aerobic exercises that includes 30 minutes (2 sets each is of 15 minutes) of treadmill, Static cycling for 15 minutes and walking for straight 20 minutes. For 7 weeks
  Interventions: Device: Glucometer
- Control Group (Self stretching) (Active Comparator): After the baseline assessment, the patient in the control group received self-stretching without aerobic exercises. Self-stretching that includes butterfly stretch, wall stretching and cat and cow pose for 5 sec each and 10 repetitions for 7 weeks
  Interventions: Device: Glucometer

INTERVENTIONS:
Device: Glucometer — A glucometer, which is a portable device used to measure blood glucose levels, was used in this study to collect data. It is a dependable and widely used tool for assessing glycemic control in people with diabetes, including gestational diabetes

SUMMARY:
: Gestational diabetes is a common pregnancy-related condition characterized by impaired glucose metabolism. It poses risks to both maternal and fetal health. Physical activity interventions, such as self-stretching and aerobic exercise, have shown potential in improving glycemic control and managing associated symptoms in individuals with diabetes. Objective: To determine the effects of self-stretching, with or without aerobic exercise, on glycemic control, fatigue, and stress for women with gestational diabetes

DETAILED DESCRIPTION:
A Randomized controlled trial was conducted at khursheed majeed Hospital Lahore and was completed in 8th month after approval of synopsis .A sample of 24 women having age 20 to 40 with gestational diabetes were selected through non probability convenience sampling technique and then randomly allocated into group A(self-stretching with aerobic exercise) and group B (self-stretching without aerobic exercise). The outcome measures were glycemic control, assessed by measuring fasting and postprandial blood glucose levels using a glucometer fatigue and stress levels, measured by Fatigue Assessment Scale (FAS) and Perceived Stress Scale (PSS), respectively. These measures will be obtained at baseline and after the 7-weeks intervention period. All participants in both groups were evaluated before and after the treatment programs.

Data was analyzed by using SPSS 25. Results: Mean value of Fasting blood glucose pre-treatment (Mean Difference=0.05) and post treatment (Mean Difference=0.14) with p value <0.05. Mean value of 2 h postprandial blood glucose pre-treatment (Mean Difference=0.04) and post treatment (Mean Difference=0.20) with p value <0.05.Mean value of Fatigue assessment scale pre-treatment (Mean Difference=1.56) and post treatment (Mean Difference=4.21) with p value <0.05. Mean value of Perceived stress scale pre-treatment (Mean Difference=1.05) and post treatment (Mean Difference=4.74) with p value <0.05 Conclusion: The study concluded that both groups Aerobic exercises + self-stretching (experimental group) and self-stretching Exercises only (control group) improve glycemic control, reduce fatigue and stress in gestational diabetes. However Aerobic exercises + self-stretching is more effective than self-stretching only

ELIGIBILITY:
Inclusion Criteria:

* Age 20 -40.
* Weight: 70kg-100kg.
* Women diagnosed with gestational diabetes.
* Second and third trimester of pregnancy

Exclusion Criteria:

* Females having history of depression
* Thyroid problems
* Preexisting diabetes • Early onset diabetes
* Multiple pregnancies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gestational Diabetes during pregnancy
Enrollment: 36 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Glucometer | 8 weeks
  A glucometer, which is a portable device used to measure blood glucose levels, was used in this study to collect data. It is a dependable and widely used tool for assessing glycemic control in people with diabetes, including gestational diabetes. These measurements provided factual information on glycemic control and help compare blood glucose levels between the self-stretching with and without aerobic exercise groups
Fatigue assessment scale | 8 weeks
  The Fatigue Assessment Scale (FAS) is a 10-item self-report scale evaluating symptoms of chronic fatigue. The FAS treats fatigue as a unidimensional construct and does not separate its measurement into different factors. However, in order to ensure that the scale evaluates all aspects of fatigue, it measures both physical and mental symptoms. This scale can be useful in tracking fatigue over time in the context of psychiatric conditions, physical illness or chronic fatigue syndrome. The FAS has an internal consistency of .90. Results on the scale also correlated highly with the fatigue-related subscales of other measures like the Checklist Individual Strength. The total score ranges from 10 to 50, with a higher score indicating more severe fatigue. A description of the fatigue experienced is presented for the total score where: less than 22 indicates "normal" (i.e. healthy) levels of fatigue, between 22 and 34 indicates mild-to-moderate fatigue and 35 or more indicates severe fatigue
Perceived stress scale: | 8 weeks
  The Perceived Stress Scale (PSS) is a classic stress assessment instrument. The tool, while originally developed in 1983, remains a popular choice for helping us understand how different situations affect our feelings and our perceived stress. The questions in this scale ask about your feelings and thoughts during the last month. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress. The Perceived Stress Scale is interesting and important because your perception of what is happening in your life is most important

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Taufiq, PPDPT, Principal Investigator — Riphah International University, Senior Lecturer
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No